CLINICAL TRIAL: NCT05490186
Title: Function, Pain, and Alignment Following Knee Replacement for the Treatment of Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely terminated due to a long pause in study activities and significant missing participant data.
Sponsor: North York General Hospital (Other)
Responsible Party: Principal Investigator, Mary Rahmat, Clinical Trials Manager, North York General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYGH REB #21-0043
Record Dates: First submitted 2021-12-07; First posted 2022-08-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Knee Replacement, Total; Pain, Postoperative; Functional Independence
MeSH Terms: conditions — Pain, Postoperative | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Manual Adjusted Mechanical Alignment (Active Comparator): Usual care:
  * Midline incision, no tourniquet, medial Parapatellar arthrotomy, resect anterior osteophytes
  * Distal femoral cut with 3-5 degrees of valgus from the anatomical axis (Based on the angle measurement on the 4 foot standing Xray). Correct for flexion contracture.
  * Measure the femoral size with the anterior referencing guides. Use 3 degrees external rotation to the Posterior condylar axis
  * Perform anterior, posterior and chamfer cuts with the 4 in 1 in appropriate external rotation
  * Extramedullary tibial alignment guide with 3-5 degrees posterior slope, and orthogonal cut to the tibial axis.
  * Resect posterior osteophytes
  * Place trial components and perform appropriate release/balance the gaps
  * Patellar replacement based on surgeon's discretion
  * Cementing the components with tourniquet inflation
  Interventions: Procedure: Total Knee Replacement
- Robotic Assisted Adjusted Mechanical Alignment (Experimental): * Midline incision, no tourniquet, medial Parapatellar arthrotomy, resect anterior osteophytes
  * Place the femoral pins in the proximal incision and the tibial pins 4 finger breadths under the joint line
  * Map the knee and perform evaluation
  * Assess gaps, adjust the femoral axis to decrease soft tissue release (+/- 2 degrees), correct for flexion contracture
  * Verify and perform distal femoral cut, proximal tibial cut orthogonal (90 Degrees) to the tibial axis
  * Assess and balance extension gap with appropriate releases
  * Remap the posterior condylar axis, assess the flexion space, 3 degrees external rotation to the posterior condylar axis
  * Perform anterior, posterior and chamber cuts with the 4 in 1 (appropriate external rotation), followed by posterior osteophyte resection
  * Place trial components and balance the knee, soft tissue releases (1-2 mm)
  * Patellar replacement based on surgeon's discretion
  * Cementing the components with tourniquet inflation
  Interventions: Procedure: Total Knee Replacement
- Robotic Assisted Kinematic Alignment: (Joint line restoration) (Experimental): -- Midline incision, no tourniquet, medial parapatellar arthrotomy, resect anterior osteophytes
  * Place femoral pins in proximal incision, tibial pins 4 finger breadths under joint line
  * Map and evaluate the knee, ROM, varus valgus testing at 0 & 90 degrees flexion
  * Distal femoral cut based on cartilage loss on medial and lateral femoral condyle (9mm total cut/condyle).
  * Perform distal femoral cut, maintain the joint line (femoral axis +/- 5 degrees)
  * Perform proximal tibial cut within +/- 3 degrees, balance the gaps, differential between medial and lateral gaps = 1- 3mm.
  * Assess extension space, resect posterior osteophytes
  * Remap posterior condylar axis, place 4 in 1 at 0 degrees to the post condylar axis (aim = 9mm posterior condylar cuts)
  * Resect posterior osteophytes, place trial components. Adjust cuts to achieve a balanced knee, maintain HKA axis +/- 3 degrees
  * Patellar replacement per surgeon discretion
  * Cement the components with tourniquet inflation
  Interventions: Procedure: Total Knee Replacement

INTERVENTIONS:
Procedure: Total Knee Replacement — Surgical technique for Total knee replacement will be standardized with a MicroPort prosthetic knee joint, patella replacement is optional based on the surgeon's assessment. The participants will receive local anesthetic infiltration by the surgeon, and a similar anesthetic technique with spinal anesthesia using epidural morphine and single shot peripheral nerve blocks. They will receive weight based antibiotics and tranexamic acid. Participants will be randomized to one of three groups. 1)Manual adjusted mechanical knee alignment (usual care) involves the surgeon manually. 2) Robot assisted surgery will include using the ROSA© device from Zimmer©. Robot assisted mechanical alignment aims for neutral alignment of the knee joint. 3) Robot assisted restricted kinematic alignment aims to place the knee joint closer to the participant's anatomical positioning.
  Other Names: Manual Adjusted Mechanical Alignment; Robotic Assisted Adjusted Mechanical Alignment; Robotic Assisted Kinematic Alignment: (Joint line restoration)

SUMMARY:
There are many factors that can influence patient satisfaction and patient related outcomes following total knee replacement including the surgical alignment of the joint components. Historically, total knee replacements have been performed with an aim aiming to achieve neutral alignment or a mechanical weight axis in the lower extremity . However, only 0.1 % of the population have a pre-surgical anatomical neutral alignment, and therefore the constitutional anatomy of the patient is neglected. There is a growing trend to return patients back their anatomical constitutional alignment after a knee replacement, referred to as Kinematic Alignment using robotics. The aim of this randomized controlled trial is to examine how mechanical alignment and kinematic alignment impacts function, pain, mood and fatigue following TKR for the treatment of osteoarthritis. Outcomes will be measured at 6 week, 6 months, 1 year and 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral TKR for the treatment of osteoarthritis
* between the age of 18 and 85 years of age
* able to read, speak and understand English, have a telephone
* are able to provide consent

Exclusion Criteria:

* enrolled in another study, are
* undergoing revision surgery or bilateral surgery, and are
* over the age of 85 years. Patients will also be excluded if they
* have a cognitive impairment (as indicated in the medical record) affecting their ability to comprehend the questions being asked

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Function | post-operatively 1 year
  Oxford knee score

SECONDARY OUTCOMES:
Quality of Life following knee surgery | post-operatively at 2 years
  EuroQol 5D index
Quality of Life following knee surgery | post-operatively at 6 weeks
  EuroQol 5D index
Quality of Life following knee surgery | post-operatively at 6 months
  EuroQol 5D index
Quality of Life following knee surgery | post-operatively at 1 year
  EuroQol 5D index
Pain intensity and effectiveness of analgesics | Post-operatively at 6 weeks
  Brief Pain Inventory-Short Form - Pain Severity Index
Pain intensity and effectiveness of analgesics | Post-operatively at 6 months
  Brief Pain Inventory-Short Form - Pain Severity Index
Pain intensity and effectiveness of analgesics | Post-operatively at 1 year
  Brief Pain Inventory-Short Form - Pain Severity Index
Pain intensity and effectiveness of analgesics | Post-operatively at 2 years
  Brief Pain Inventory-Short Form - Pain Severity Index
Satisfaction with knee surgery | Post-operatively at 6 weeks, 6 months, 1 year and 2 years
  Forgotten Joint Score
Satisfaction with knee surgery | Post-operatively at 6 weeks
  Forgotten Joint Score
Satisfaction with knee surgery | Post-operatively at 6 months
  Forgotten Joint Score
Satisfaction with knee surgery | Post-operatively at 1 year
  Forgotten Joint Score
Satisfaction with knee surgery | Post-operatively at 2 years
  Forgotten Joint Score
Function | post-operatively at 6 weeks
  Oxford knee score
Function | post-operatively at 6 months
  Oxford knee score
Function | pre-operatively
  Oxford knee score
Function | post-operatively at 2 years
  Oxford knee score

OTHER OUTCOMES:
Health Care Utilization | Post-operatively at 6 weeks
  unanticipated visits to emergency department, primary care provide, surgeon due to knee surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frank Mastrogiacomo, PhD, Principal Investigator — North York General Hospital
Locations (1):
- North York General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Knowledge translation will occur utilizing a variety of mechanisms. The results of this study will be disseminated at the Canadian Orthopaedic Association conference. They will also be published in an high impact journal. At the provincial level, the data from this study will be shared with Health Quality Ontario, as a requirement of the bundled care program. At the local level, the investigators will disseminate the results of this study as aggregate data at North York General Hospital with to the health care practitioners and administrators involved with caring for the arthroplasty patient population.